CLINICAL TRIAL: NCT01085981
Title: The Quantitative Analysis of Clitoral Blood Before and After a Topically Applied Vasodilating Cream Using Sonographic Doppler Flow Plethysmography
Brief Title: Assessing the Effects of a Topically Applied Cream to Clitoral Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: East Suburban Ob Gyn (Other)
Responsible Party: michael pelekanos md, East suburban OBGYN
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-006
Record Dates: First submitted 2010-03-02; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Female Sexual Dysfunction
Keywords: quantitative assessment of the effects of a topically; applied vasodilating cream to the clitoris using doppler; flow plethysmography
MeSH Terms: interventions — Arginine; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GRAS ingredients cream (Active Comparator): The study will be placebo controlled double blind study which will require two office visits after informed consent and sensitivity testing done with the study cream on the day of recruitment.
  On the first office visit the patient will have their baseline clitoral and uterine blood flow measured quantitatively by the same sonographer using the General electric Voluson 700 unit Then placebo or active cream will be applied and the pt restudied. the same process is repeated another day with the second arm cream.
  Interventions: Drug: arginine 20%, nicotinamide .01%, niacin.1%, in LipodermPG 50%; Drug: GRAS cream
- placebo cream then doppler study (Placebo Comparator)
  Interventions: Drug: arginine 20%, nicotinamide .01%, niacin.1%, in LipodermPG 50%; Drug: Topical study cream

INTERVENTIONS:
Drug: arginine 20%, nicotinamide .01%, niacin.1%, in LipodermPG 50% — On the first office visit the patient will have their baseline clitoral and uterine blood flow measured quantitatively by the same sonographer using the General electric Voluson 700 unit. Clitoral blood flow will be accessed utilizing the 12 megahertz linear probe. With light pressure, the probe will be applied sagittally and proximal to the clitoral hood with an angle less than 20 degrees. Peak clitoral artery systolic and end diastolic velocity will be measured and resistive index values will be recorded. Then utilizing the 7.5 megahertz vaginal probe baseline uterine artery flow measurements will also be obtained and recorded. With both GRAS cream and placebo.
  Other Names: Temptation tc
Drug: Topical study cream — One gram applied to clitoris by nurse then ten minutes later doppler study of clitoral blood flow
  Other Names: Temptation tc
  Arms: placebo cream then doppler study
Drug: GRAS cream — 1 gram of active cream will be applied by nurse then 10 minutes later clitoral blood flow will be assessed by doppler studies see protocol
  Other Names: Temptation tc
  Arms: GRAS ingredients cream

SUMMARY:
The purpose of this study is to determine if blood flow to the clitoris is increased by topically applying a cream that causes increased blood flow. This will be measured with a sonogram.

DETAILED DESCRIPTION:
On the first office visit the patient will have their baseline clitoral and uterine blood flow measured quantitatively by the same sonographer using the General electric Voluson 700 unit. Clitoral blood flow will be accessed utilizing the 12 megahertz linear probe. With light pressure, the probe will be applied sagittally and proximal to the clitoral hood with an angle less than 20 degrees. Peak clitoral artery systolic and end diastolic velocity will be measured and resistive index values will be recorded. Then utilizing the 7.5 megahertz vaginal probe baseline uterine artery flow measurements will also be obtained and recorded.

The patient will then be placed in an exam room and the same nurse practitioner will apply the GRAS cream or the placebo to the patients' clitoral hood with minimal manipulation. Ten minutes later the sonographer will repeat the two scans and record the same measurements as before. The patient will then come back another day to repeat the above process. Patients will be coded to assure that which ever cream they received the first visit they will get the opposite the second time. The creams will be blinded to the nurse practitioner, the patient, the sonographer, and the principle investigator.

GRAS cream is arginine 20%, nicotinamide .01%, niacin.1%, in LipodermPG 50%,

ELIGIBILITY:
Inclusion Criteria:

* Healthy sexually active females ages 25-60 years

Exclusion Criteria:

* Not eligible if they are experiencing sexual pain disorders
* Psychological sexual aversion disorders
* Vaginismus
* Pregnant/nursing
* Diabetes mellitus
* Central nervous system disorders
* Psychosis
* Currently on any SSRI's, or any other condition that may effect the patient from reliably signing the informed consent.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
to determine the effect study cream has on clitoral blood flow | ten minutes after application of active or placebo
  the blood flow analysis will be measured with doppler flow plethysmography

SECONDARY OUTCOMES:
to determine the effect study cream has on uterine blood flow | measuring uterine flow with doppler 10 minutes after application
  see previous description

CONTACTS AND LOCATIONS:
Overall Officials: michael j pelekanos, md, Principal Investigator — east suburban obgyn
Locations (1):
- East Suburban Obgyn, Monroeville, Pennsylvania, United States